CLINICAL TRIAL: NCT04741347
Title: Transverse Fractures +/- Posterior Wall of the Acetabulum: Predictors of the Quality of Surgical Reduction and Long-term Outcome
Brief Title: Predictors of the Quality of Surgical Reduction and Long-term Outcome
Acronym: Fracture_Trans
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Fracture_Trans
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-09

CONDITIONS: Transverse Fracture of Acetabulum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acetabulum fractures are complex, relatively rare lesions linked to a more or less good functional prognosis and therefore represent a real surgical challenge.

In the literature, it is accepted that surgical delay, among other things, negatively impacts the quality of surgical reduction. However, this reduction must be a major priority since it is one of the factors conditioning the functional result.

In our study, we wish to analyze a particular type of fracture, less studied, or with small series, that are the transverse fractures (+/- posterior wall), known for their difficulty of reduction. The reduction is even greater as the fracture line often passes through the acetabular bearing zone, compromising the functional prognosis.

The choice of surgical approach for this type of fracture is controversial. More and more, a single approach, usually posterior, without compulsory fixation of the anterior component of the transverse fracture is preferred over the traditional double approach anterior and posterior, and this in particular to reduce the morbidity of this surgery.

But this one-size-fits-all approach does not always achieve a good reduction and it is believed that the time to surgery may play a role.

If it is accepted that the surgical delay before reduction in osteosynthesis of an acetabular fracture is involved in the quality of the reduction and therefore the functional result in these patients, the question asked is whether this delay should condition the choice of a double approach, anterior and posterior, for this type of fracture (transverse +/- posterior wall).

Indeed, with increasing surgical time, the risk of scar tissue formation and early callus increases, making bone fragments less mobile, reduction more difficult and indirect reduction techniques (which are used when single approach is chosen) less efficient.

In addition, most of the studies evaluating the quality of reduction of acetabular fractures use a radiographic score, that of Matta.

However, it has been shown that the CT scan was more efficient than the x-rays in detecting a residual displacement of the fracture. Also, in this study, we want to analyze the quality of reduction thanks to the scanner, which is rarely done in the literature.

This work aims to determine the predictive factors of the quality of reduction of transverse fractures +/- posterior wall of the acetabulum, evaluated on the postoperative CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with transverse fractures +/- posterior wall of the acetabulum
* Patient cared for at Paris Saint-Joseph Hospital, between 2006 and 2020
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient under legal protection
* Patient deprived of liberty
* Patient not operated
* Patient with an undisplaced fracture
* Patient who did not have a post-operative control scan
* Patient objecting to the use of their data for this research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were treated for transverse fractures +/- posterior wall of the acetabulum within the Paris Saint-Joseph Hospital Group, between 2006 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Fracture reduction quality | Year 1
  This outcome corresponds to the fracture reduction quality assessed on the postoperative CT scan using the Saint Joseph score.

SECONDARY OUTCOMES:
Complication rate | Year 1
  This outcome corresponds to the rate of postoperative complications (infection, hematoma, anemia requiring transfusion, neurological complications (e.g. sciatic nerve injury)).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume RIOUALLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Matta JM. Fractures of the acetabulum: accuracy of reduction and clinical results in patients managed operatively within three weeks after the injury. J Bone Joint Surg Am. 1996 Nov;78(11):1632-45. PMID 8934477
- [Result] Madhu R, Kotnis R, Al-Mousawi A, Barlow N, Deo S, Worlock P, Willett K. Outcome of surgery for reconstruction of fractures of the acetabulum. The time dependent effect of delay. J Bone Joint Surg Br. 2006 Sep;88(9):1197-203. doi: 10.1302/0301-620X.88B9.17588. PMID 16943472
- [Result] Giordano V, do Amaral NP, Pallottino A, Pires e Albuquerque R, Franklin CE, Labronici PJ. Operative treatment of transverse acetabular fractures: is it really necessary to fix both columns? Int J Med Sci. 2009 Jul 12;6(4):192-9. doi: 10.7150/ijms.6.192. PMID 19652723
- [Result] Verbeek DO, van der List JP, Villa JC, Wellman DS, Helfet DL. Postoperative CT Is Superior for Acetabular Fracture Reduction Assessment and Reliably Predicts Hip Survivorship. J Bone Joint Surg Am. 2017 Oct 18;99(20):1745-1752. doi: 10.2106/JBJS.16.01446. PMID 29040129